CLINICAL TRIAL: NCT00513825
Title: The Evaluation of the Effect of Sodium Bicarbonate Solution in Decreasing the Incidence of Contrast Induced Nephropathy (CIN) in Patients With Pulmonary Edema,Severe Heart Failure or Uncontrolled Hypertension
Brief Title: Preventing Contrast Nephropathy With Sodium Bicarbonate in Patients With Pulmonary Edema,Heart Failure,Uncontrolled HTN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Tehran Heart Center (Other)
Responsible Party: Ali Vasheghani Farahani, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 85-02-30-3595(2)
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2008-11-26 (Estimated); Status verified 2008-11

CONDITIONS: Contrast Induced Nephropathy
Keywords: Contrast Nephropathy; Sodium Bicarbonate; Prevention
MeSH Terms: interventions — Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 1075 cc of 77 mEq/L solution of NaCl 0.45% , prepared by adding 75 cc of 77 mEq/L NaCl 0.45 % to 1000 cc of 77 mEq/L NaCl 0.45%
  Interventions: Drug: Sodium Bicarbonate
- 2 (Active Comparator): 1075 cc fluid made by adding 75 cc of sodium bicarbonate solution 8.4% to 1000 cc of NaCl 0.45%.
  Interventions: Drug: Sodium Bicarbonate

INTERVENTIONS:
Drug: Sodium Bicarbonate — IV solution of NaCl 0.45% (Arm 1) or IV 75 cc of sodium bicarbonate 8.4% solved in 1 liter of NaCl 0.45% (Arm 2) . Each fluid is infused at the rate of 3 ml/kg/ hour one hour before the angiographic procedure, continuing at the rate of 1 ml/kg/ hour for 6 hours after the procedure. Maximum rate of fluid permitted is that for a body weight of 110 Kg.

SUMMARY:
Radio Contrast Induced Nephropathy (RCIN) remains a well recognized complication in patients undergoing diagnostic or interventional procedures requiring radiographic contrast agents. Recent studies have shown benefit in administering Sodium Bicarbonate over normal saline( the uniformly accepted prophylaxy) in preventing RCIN.But most studies have excluded patients with history of pulmonary edema, severe heart failure(NYHA 3-4), uncontrolled hypertension or ejection fraction less than 30%. Therefore the aim of this study is to evaluate the efficacy of sodium bicarbonate solved in half saline compared with infusion of half saline in prevention of RCIN in these groups of patients.

DETAILED DESCRIPTION:
Radio Contrast Induced Nephropathy (RCIN) remains a well recognized complication in patients undergoing diagnostic or interventional procedures requiring radiographic contrast agents and is the third leading cause of acquired acute renal failure in hospitalized patients. Strategies for the prevention of radiocontrast nephropathy have focused on countering vasoconstriction (pre-hydration, fenoldopam, and theophylline), enhancing flow through the nephron (diuretics), or protection against oxygen-free-radical injury (urinary alkalinization and N-acetylcysteine).

Among all prophylactic measures that have been proposed, adequate preprocedural and postprocedural hydration has demonstrated effectiveness in the prevention of radiocontrast nephropathy. Thus, it remains the most frequently applied measure in clinical practice.

A Recent study in May 2004 have shown benefit in administering Sodium Bicarbonate over normal saline as a prophylaxy.Since alkalizing renal tubular fluid with bicarbonate may reduce injury .

Most studies have excluded patients with history of pulmonary edema, severe heart failure(NYHA 3-4), uncontrolled hypertension or ejection fraction less than 30% and no specific protocol is tested for this group of patients. This study focuses on preventing RCIN in this specific group of patients .

Comparisons:1075 cc NaCl 0.45% or 75 cc of sodium bicarbonate 8.4% solved in one liter of NaCl 0.45%. Each fluid is infused at the rate of 3 ml/kg/ hour one hour before the angiographic procedure, continuing at the rate of 1 ml/kg/ hour for 6 hours after the procedure. Maximum rate of fluid permitted is that for a body weight of 110 Kg.

ELIGIBILITY:
Inclusion Criteria:

* individuals aged 18 years or older with serum creatinine levels of at least 1.5 mg/dl , who were scheduled to undergo diagnostic or therapeutic coronary artery angiography.
* Patients with a history of Pulmonary edema or
* Patients with severe Heart Failure ( NYHA 3-4) or
* Patients with ejection fraction of less than 30% on Echocardiography ( done in the previous month of admission) or
* Patients with uncontrolled hypertension (treated systolic blood pressure more than 160 mmHg, or diastolic blood pressure more than 100mmHg )

Exclusion Criteria:

* serum creatinine levels of more than 8 mg/dl
* previous history of dialysis
* GFR < 20 ( as calculated with this formula: ((140-Age)(Weight(Kg)) / Serum Creatinine(mg/dl) ×72 ) , in females GFR was multiplied by 0.85 )
* emergency catheterization
* recent exposure to radiographic contrast agents (within previous two days of the study)
* radiocontrast agent dosage needed more than 300 gr during the procedure
* allergy to radiocontrast agent
* pregnancy
* administration of dopamine, mannitol , fenoldopam or N-Acetyl Cystein during the intended time of study
* need for continuous hydration therapy (e.g. sepsis )
* history of Multiple myeloma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2007-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
development of contrast induced nephropathy defined as an absolute (> or = 0.5 mg/dl) or relative increase (> or = 25%) in serum creatinine at 48 hours after exposure to a contrast agent compared to baseline serum creatinine values. | at 48 hours

SECONDARY OUTCOMES:
an absolute (> or = 0.5 mg/dl) or relative increase(> or= 25% ) in serum creatinine at day 5 after exposure to a contrast agent. | at day 5
Urine PH after initial bolus | within 6 hours after initial bolus
development of contrast induced nephropathy defined as 25% decrease in glomerular filtration rate (GFR) at 48 hours. | at 48 hours
development of contrast induced nephropathy defined as 25% decrease in glomerular filtration rate (GFR)on day 5 . | on day 5 post contrast

CONTACTS AND LOCATIONS:
Overall Officials: Ali Farahani Vasheghani, M.D., Study Director — Tehran University of Medical Sciences, Tehran Heart Center; Ebrahim Kassaian, M.D., Principal Investigator — Tehran Heart Center; Akbar Fotuhi, M.D., Principal Investigator — Tehran Heart Center; Mohammad Reza Khatami, M.D., Principal Investigator — Tehran Heart Center; Mojtaba Salarifar, M.D., Principal Investigator — Tehran Heart Center; Ebrahim Nematipur, M.D., Principal Investigator — Tehran Heart Center; Ahmad Iaminisharif, M.D., Principal Investigator — Tehran Heart Center; Saeid Sadeghian, M.D., Principal Investigator — Tehran Heart Center; Ali mohammad Hajzeinali, M.D., Principal Investigator — Tehran Heart Center; Mohammad Alidoosti, M.D., Principal Investigator — Tehran Heart Center; Hamidreza Purhosseini,, M.D., Principal Investigator — Tehran Heart Center; Ali Kazemisaeid, M.D., Principal Investigator — Tehran Heart Center; Gholamreza Davoodi, M.D., Principal Investigator — Tehran Heart Center; Alireza Amirzadegan, M.D., Principal Investigator — Tehran Heart Center; Abbas Soleimani, M.D., Principal Investigator — Tehran Heart Center; Sirus Darabian, M.D., Principal Investigator — Tehran Heart Center; Kianush Hossein, M.D., Principal Investigator — Tehran Heart Center; Gelareh Sadigh, M.D., Principal Investigator — Tehran University of Medical Sciences; Amir Hossein Razavi, M.D., Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Tehran Heart Center, Tehran, Iran